CLINICAL TRIAL: NCT04061694
Title: Immediate Loading of Single Implants, Guided Surgery, Digital Impression and CAD/CAM Technology: Clinical and Patient-centered Outcome.
Brief Title: Immediate Loading and Fully Guided Surgery: Single Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Folktandvården Skåne AB (Other)
Responsible Party: Principal Investigator, Björn Gjelvold, Specialist in Oral Prosthodontics, Folktandvården Skåne AB
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIL001
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Osseointegration Failure of Dental Implant
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Immediate loading (Experimental): Single dental implant installed with the assistance of fully guided-surgery, submitted to immediate loading with restorations fabricated with the help of intraoral scanning and 3D printing
  Interventions: Procedure: Immediate loading, fully guided surgery and 3D printed restoration
- Immediate loading (Other): Historic cohort subjected to immediate loading
  Interventions: Procedure: Immediate loading

INTERVENTIONS:
Procedure: Immediate loading, fully guided surgery and 3D printed restoration — Fully guided surgery installation of single dental implants. 3D printed restorations that were immediate loaded.
  Arms: Digital Immediate loading
Procedure: Immediate loading — Only subjected to immediate loading. Conventional procedure.
  Arms: Immediate loading

SUMMARY:
To evaluate the overall treatment outcome of single implants installed with the assistance of fully guided-surgery, submitted to immediate loading with restorations fabricated with the help of intraoral scanning, during a 1-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age who had signed an informed consent
* in need of a single-tooth replacement of an incisor, canine or pre-molar in the maxilla.

Exclusion Criteria:

* general contraindications for oral surgery
* patients with inadequate oral hygiene
* need for bone grafting or ridge augmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Wennerberg, PhD, Study Director — Göteborg University
Locations (1):
- Centre of Dental Specialist Care, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Immediate Loading | Immediate Loading
Started | 21 | 25
Completed | 19 | 25
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Immediate Loading | Immediate Loading | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (21.0) | 40.8 (13.3) | 40.5 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Implant Survival
Description: Survival of dental implants. Implant survival means that implants are still in the mouth at the time of examination, regardless of the state of the prosthesis or patient satisfaction
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Digital Immediate Loading | Immediate Loading
Number analyzed (Participants) | 21 | 25
participants | 19 | 25

2. Primary Outcome: MBL
Description: Marginal bone loss MBL, measured in mm from implant abutment junction.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Digital Immediate Loading | Immediate Loading
Number analyzed (Participants) | 19 | 25
mm | -0.40 (0.41) | -0.57 (0.52)

3. Primary Outcome: Pink Esthetic Score
Description: Pink Esthetic Score (PES) Soft-tissue aesthetic scale. Range 0-14. Min = 0, aesthetic failure. Max = 14, almost prefect aesthetic outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Immediate Loading | Immediate Loading
Number analyzed (Participants) | 19 | 25
score on a scale | 10.53 (2.04) | 10.36 (2.46)

4. Primary Outcome: White Esthetic Score
Description: White Esthetic Score (WES) Dental crown/tooth aesthetic scale. Range 0-10. Min = 0, aesthetic failure. Max = 10, almost prefect aesthetic outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Immediate Loading | Immediate Loading
Number analyzed (Participants) | 19 | 25
score on a scale | 7.79 (1.36) | 7.76 (1.30)

5. Primary Outcome: Oral Health Impact Profile - 14
Description: Oral health impact profile - 14 (OHIP-14) Oral health related quality of life questioner. Score range 14-70. Low score indication good oral health related quality of life. High score indicates the opposite.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Immediate Loading | Immediate Loading
Number analyzed (Participants) | 19 | 25
score on a scale | 17.10 (3.23) | 16.48 (3.87)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious events: loss of dental implant. Other adverse event: prosthetic restoration complications.
Arm/Group | Digital Immediate Loading | Immediate Loading
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/25
Other Adverse Events (participants affected / at risk) | 0/21 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Digital Immediate Loading (N=21) | Immediate Loading (N=25)
Dental implant loss (Surgical and medical procedures) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04061694/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04061694/SAP_001.pdf